CLINICAL TRIAL: NCT06338319
Title: Book Sharing for Toddlers With Clefts
Acronym: BOOST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); Nationwide Children's Hospital (Other); Children's Hospital Los Angeles (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-048-E
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cleft Palate; Cleft Lip and Palate
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BOOST Program (Experimental): Parents in the BOOST Program group will receive books to read with their children and send smartphone video recordings of their reading interactions.
  To provide support, parents will participate in 3 remote, parent-focused book-sharing intervention sessions
  Interventions: Behavioral: Book-Sharing for Toddlers with Clefts (BOOST)
- Standard of Care Comparison Group (No Intervention): Parents in the Standard of Care Comparison Group will receive books to read with their children and send smartphone video recordings of their reading interactions.
  Parents in the comparison group will not participate in BOOST intervention sessions.

INTERVENTIONS:
Behavioral: Book-Sharing for Toddlers with Clefts (BOOST) — BOOST is a dialogic book-sharing intervention. Topics covered include strategies to increase the frequency of shared reading, child engagement and involvement in reading, and strategies to promote language development. Handouts will be shared during the sessions (using the Zoom share screen feature) and sent to families to summarize the content. Parents will record and securely upload shared reading videos during the intervention period. The research team will send prompts for these video uploads after each intervention session. Interventionists will review these videos between sessions to identify parent strengths, application of target skills, and opportunities for improvement.
  Arms: BOOST Program

SUMMARY:
Children with clefts exhibit difficulty with language and literacy compared to children without clefts. However, little is known about interventions to address these difficulties in the cleft population. This study will test the efficacy of a parent-focused dialogic book-sharing intervention for toddlers with isolated cleft palate. The study will use a randomized controlled trial (RCT) design and Intention to Treat (ITT) analyses. Child outcomes include expressive and receptive language. Parent outcomes of interest include the frequency and quality of shared reading interactions. To assess mechanisms of action, the study will test whether changes in child outcomes are mediated by changes in parents' behavior. Analyses will also explore heterogeneity in outcomes to determine whether the intervention is more effective in certain clinical or demographic sub-groups.

ELIGIBILITY:
Inclusion Criteria:

* A child's parent or primary caregiver provides a signed and dated informed consent form and permission for their child to participate.
* A child's parent is willing to comply with all study procedures and be available for the duration of the study.
* Child is between the ages of 20 to 32 months at the time of enrollment.
* Child has been diagnosed with isolated cleft palate, with or without cleft lip.
* Child has received palate repair surgery.
* The family's preferred language is English or Spanish.
* The family has access to a smartphone or similar device (e.g., tablets) capable of recording and sending videos.

Exclusion Criteria:

* Diagnosed genetic condition associated with developmental delay (e.g., 22q11 deletion).
* The child has a diagnosis of autism spectrum disorder
* The child has a tracheostomy tube
* Child delivered < 32 weeks' gestation.
* Child in state custody or foster care.
* Child with significant sensory impairment (blindness, sensorineural hearing loss).
* The caregiver speaks a language other than English or Spanish
* The caregiver does not own a smartphone or similar device capable of recording/sending video

Ages: 20 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Expressive One Word Picture Vocabulary Test-Fourth Edition | End of study (At least 8 weeks after the end of the intervention period)
  Standardized, clinician-administered measure of expressive language. Possible raw scores range from 0 to 190, with higher scores indicating better expressive language
Receptive One Word Picture Vocabulary Test-Fourth Edition | End of study (At least 8 weeks after the end of the intervention period)
  Standardized, clinician-administered measure of receptive language. Raw scores range from 0 to 190, with higher scores indicating better receptive language.
Child Language Sample | End of study (At least 8 weeks after the end of the intervention period)
  Observational measure to assess child expressive language. We will obtain a count of the number of clear and intelligible utterances, the number of unique words used, and mean length of utterance. Higher scores indicate better child language skills.
MacArthur-Bates Communicative Development Inventory - Computer Adaptive Test | Baseline and at end of study (at least 8 weeks after the end of the intervention period)
  Parent report measure of children's expressive language. Raw scores range from 0 to 50, with higher scores indicating better expressive language.

SECONDARY OUTCOMES:
Child Speech Sample - Percent Consonants Correct - Revised, Total Number of Unique Consonants | Baseline and at end of study (at least 8 weeks after the end of the intervention period)
  Parent-administered measure to assess children's speech sound inventory and production accuracy. Children will be asked to name approximately 27 pictures. Responses will be recorded and phonetically transcribed to obtain a count of consonant sounds attempted and consonant sounds correct in the beginning, middle, and final positions for the pictured words. We will use these counts to obtain percent consonants correct - revised (#consonants correct/#consonants attempted). Higher scores indicate better speech sound accuracy. We will also count the total number of unique consonants produced, with higher scores indicating larger phonetic inventory.

OTHER OUTCOMES:
Frequency of Shared Reading | Throughout the intervention period of approximately 8 weeks and again at end of study (at least 8 weeks after the end of the intervention period)
  Parent report measure of shared reading, reported as the number of books read with their child in the last 24-hours. Higher scores indicate more frequent shared reading.
Quality of Shared Reading | Throughout the intervention period of approximately 8 weeks and again at end of study (at least 8 weeks after the end of the intervention period)
  Observational measure of parent-child reading interactions, including a count of the dialogic book-sharing strategies used during the observation. Higher scores indicate higher quality shared reading interaction.
Child Language During Reading | Throughout the intervention period of approximately 8 weeks and again at end of study (at least 8 weeks after the end of the intervention period)
  Observation of child language during reading interactions, including a count of the number of clear and intelligible utterances the child uses, the number of unique words, and the mean length of utterance. Higher scores will indicate better observed child language skills.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Collett, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No